CLINICAL TRIAL: NCT00623740
Title: Early Prevention of Broncho-pulmonary Dysplasia and Neonatal Mortality in Very Preterm Infants Using Low Dose of Hydrocortisone: a Randomized Controlled Trial
Brief Title: PREMILOC Trial to Prevent Bronchopulmonary Dysplasia in Very Preterm Neonates
Acronym: PREMILOC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P 060250; 2007-002041-20 (EudraCT Number)
Record Dates: First submitted 2008-02-07; First posted 2008-02-26 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2016-08

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: Hydrocortisone; Very low birth weight; Bronchopulmonary dysplasia; Prevention Cerebral palsy
MeSH Terms: conditions — Bronchopulmonary Dysplasia | interventions — Hydrocortisone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1: hydrocortisone (Experimental): 1: active arm treated with low doses of HC during the first 10 days of life
  Interventions: Drug: hydrocortisone
- 2: Placebo (Placebo Comparator): 2:placebo arm treated with placebo at the same conditions than active arm
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: hydrocortisone — Intravenous slow of hemisuccinate hydrocortisone 0.5 mg/kg/12 hours during 7 days then 0.5mg/kg/24 hours during 3 days.
  Other Names: hydrocortisone upjohn 100mg
  Arms: 1: hydrocortisone
Drug: placebo — intravenous slow of placebo 0.5mg/kg/12 hours during 7 days then 0.5 mg/kg/24 hours during 3 days
  Arms: 2: Placebo

SUMMARY:
There is increasing evidence linking a fetal and early neonatal systemic inflammatory response syndrome to the subsequent development of bronchopulmonary dysplasia (BPD) and white matter injury (WMI) in very preterm infants. Babies with evidence of adrenal insufficiency early in life may not be able to control the inflammatory response and are thereby more likely to develop BPD than babies who do not show such evidence of inflammation. We designed a randomized controlled trial to test the hypothesis whether very preterm babies at high-risk of BPD, treated with low doses of HC during the first 10 days of life, are more likely to survive without BPD at 36 weeks of post-menstrual age (PMA), compared to babies treated with placebo.

DETAILED DESCRIPTION:
Individual patients and study procedures. Entry criteria: gestational age between 24 weeks and 27 weeks + 6 days, babies born to mother with either clinical chorioamnionitis, preterm and prelabor rupture of the membranes (PPROM), or preterm labor, written informed consent obtained before inclusion and randomization. Exclusion criteria: babies born with birth weight below the 3th percentile, PPROM before 22 weeks, major fetal anomaly or congenital malformation, mother refusal or inability to provide consent. Stratification: stratum A: 24-25 weeks and stratum B: 26-27 weeks. Centrally controlled randomization takes place between 12 and 48 hours of age and patients assigned to the HC group are treated with 0,5 mg/kg HC intravenously twice a day for seven days and once a day for the next three days. Ibuprofen is only given to babies with persistent ductus arteriosis (PDA) echocardiographically confirmed at 24 hours of age or older.

Outcome variables. The primary outcome is a dichotomous variable: survival without BPD at 36 weeks PMA. A consistent physiologic definition of BPD will be used by all participating centres (Walsh MC, Pediatrics 2004;114:1305-11). Secondary outcome variables include features of WMI on MRI performed at 40 weeks PMA and neurodevelopmental outcome at 2-year of corrected age. Other outcome variables include death before discharge, BPD at 28 days and 36 weeks, duration of mechanical ventilation and O2 supplementation, need for vasopressors, use of open-labeled postnatal steroids (HC or dexamethasone), confirmed or suspected early and late onset sepsis, PDA, gastrointestinal perforation, NEC, ROP, IVH, biological markers of the neonatal inflammatory response syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age between 24 weeks and 27 weeks + 6 days
* Babies born to mother with either clinical chorioamnionitis, preterm and prelabor rupture of the membranes (PPROM), or preterm labor
* Written informed consent obtained before inclusion and randomization.

Exclusion Criteria:

* Babies born to mothers with birth weight below the 3th percentile
* PPROM before 22 weeks
* Major fetal anomaly or congenital malformation
* Mother refusal or inability to provide consent.

Max Age: 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 523 (Actual)
Dates: Start 2008-04; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
dichotomous variable: survival without BPD at 36 weeks PMA. | add 8 to12

SECONDARY OUTCOMES:
features of WMI on MRI performed between 36-40 weeks PMA | 8-12 weeks
neurodevelopmental outcome | 18 month-3 years
Death before discharge | discharge
BPD 28 days and 36 weeks | 28 days and 36 weeks
duration of mechanical ventilation and O2 supplementation | inclusion to discharge
need for vasopressors | inclusion to discharge

CONTACTS AND LOCATIONS:
Overall Officials: olivier BAUD, Pr, Principal Investigator — ASSISTANCE PULIQUE HOPITAUX DE PARIS
Locations (1):
- Hopital Robert Debre, Paris, France

REFERENCES:
- [Result] Baud O. [Postnatal steroid treatment in preterm infants: risk/benefit ratio]. J Gynecol Obstet Biol Reprod (Paris). 2005 Feb;34(1 Suppl):S118-26. doi: 10.1016/s0368-2315(05)82698-5. French. PMID 15767942
- [Result] Baud O, Maury L, Lebail F, Ramful D, El Moussawi F, Nicaise C, Zupan-Simunek V, Coursol A, Beuchee A, Bolot P, Andrini P, Mohamed D, Alberti C; PREMILOC trial study group. Effect of early low-dose hydrocortisone on survival without bronchopulmonary dysplasia in extremely preterm infants (PREMILOC): a double-blind, placebo-controlled, multicentre, randomised trial. Lancet. 2016 Apr 30;387(10030):1827-36. doi: 10.1016/S0140-6736(16)00202-6. Epub 2016 Feb 23. PMID 26916176
- [Result] Baud O, Trousson C, Biran V, Leroy E, Mohamed D, Alberti C; PREMILOC Trial Group. Association Between Early Low-Dose Hydrocortisone Therapy in Extremely Preterm Neonates and Neurodevelopmental Outcomes at 2 Years of Age. JAMA. 2017 Apr 4;317(13):1329-1337. doi: 10.1001/jama.2017.2692. PMID 28384828
- [Result] Baud O, Alberti C, Mohamed D, Watterberg K. Low-dose hydrocortisone in extremely preterm infants - Authors' reply. Lancet. 2016 Sep 17;388(10050):1158-9. doi: 10.1016/S0140-6736(16)31611-7. Epub 2016 Sep 16. No abstract available. PMID 27650090
- [Derived] Baud O, Lehert P; PREMILOC study group. Prophylactic hydrocortisone and the risk of sepsis in neonates born extremely preterm. Eur J Pediatr. 2025 Jun 14;184(7):419. doi: 10.1007/s00431-025-06248-9. PMID 40515786
- [Derived] Baud O, Lehert P; PREMILOC study group. Bronchopulmonary dysplasia to predict neurodevelopmental impairment in infants born extremely preterm. Pediatr Res. 2025 Jun;97(7):2436-2442. doi: 10.1038/s41390-024-03601-w. Epub 2024 Oct 24. PMID 39448816
- [Derived] Baud O, Lehert P; PREMILOC study group. The beneficial effect of prophylactic hydrocortisone treatment in extremely preterm infants improves upon adjustment of the baseline characteristics. Pediatr Res. 2024 Jan;95(1):251-256. doi: 10.1038/s41390-023-02785-x. Epub 2023 Aug 31. PMID 37653218
- [Derived] Trousson C, Toumazi A, Bourmaud A, Biran V, Baud O. Neurocognitive outcomes at age 5 years after prophylactic hydrocortisone in infants born extremely preterm. Dev Med Child Neurol. 2023 Jul;65(7):926-932. doi: 10.1111/dmcn.15470. Epub 2022 Nov 23. PMID 36417367
- [Derived] Renolleau C, Toumazi A, Bourmaud A, Benoist JF, Chevenne D, Mohamed D, Alberti C, Biran V, Baud O; PREMILOC Trial Study Group. Association between Baseline Cortisol Serum Concentrations and the Effect of Prophylactic Hydrocortisone in Extremely Preterm Infants. J Pediatr. 2021 Jul;234:65-70.e3. doi: 10.1016/j.jpeds.2020.12.057. Epub 2020 Dec 24. PMID 33359303
- [Derived] Alison M, Tilea B, Toumazi A, Biran V, Mohamed D, Alberti C, Bourmaud A, Baud O; PREMILOC Trial group. Prophylactic hydrocortisone in extremely preterm infants and brain MRI abnormality. Arch Dis Child Fetal Neonatal Ed. 2020 Sep;105(5):520-525. doi: 10.1136/archdischild-2019-317720. Epub 2020 Jan 24. PMID 31980445
- [Derived] Heneau A, Guimiot F, Mohamed D, Rideau Batista Novais A, Alberti C, Baud O; PREMILOC Trial study group. Placental Findings and Effect of Prophylactic Hydrocortisone in Extremely Preterm Infants. Pediatrics. 2018 Feb;141(2):e20171788. doi: 10.1542/peds.2017-1788. Epub 2018 Jan 18. PMID 29348196